CLINICAL TRIAL: NCT03398395
Title: Comparison of Long Term Clinical Efficacy of Different Computer-Aided Design & Computer-Aided Manufacturing(CAD/CAM) Materials for the Restoration of Teeth With Root Canal Therapy With Endocrown or 90° Shoulder Endocrown
Brief Title: Endocrown and 90° Shoulder Endocrown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2017-141
Record Dates: First submitted 2017-12-28; First posted 2018-01-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Endocrown Restoration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endocrown restoration (Active Comparator): a cervical margin in the form of a butt joint and a preparation of the pulp chamber that does not extend into the root canals.
  Interventions: Procedure: endocrown restoration
- 90° shoulder endocrown restoration (Active Comparator): a 90°cervical margin in the form of a butt joint and a preparation of the pulp chamber that does not extend into the root canals.
  Interventions: Procedure: 90° shoulder endocrown restoration

INTERVENTIONS:
Procedure: endocrown restoration — a cervical margin in the form of a butt joint and a preparation of the pulp chamber that does not extend into the root canals.
  Arms: endocrown restoration
Procedure: 90° shoulder endocrown restoration — a 90°cervical margin in the form of a butt joint and a preparation of the pulp chamber that does not extend into the root canals.
  Arms: 90° shoulder endocrown restoration

SUMMARY:
Use chairside Computer-Aided Design & Computer-Aided Manufacturing(CAD/CAM) system (computer aided design / manufacture), using glass ceramic zirconia enhanced lithium silicate glass ceramics (VITA, SUPRINITY, VS) material, compare the difference of firmness, comfort and durability between two kinds of root canal restoration methods:endocrown and 90° shoulder endocrown. Objective to establish the optimal method and material for the restoration of the teeth with root canal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 year old patients with healthy body, the tooth is molar, root tip no obvious damage, no root fracture by X-ray;
2. after complete root canal therapy, the remaining 4 wall intact tooth tissue;
3. after complete root canal therapy, the remaining 3 wall intact tooth tissue;
4. have good oral hygiene habits;
5. agreed to participate in the trial and signed the informed consent form;
6. patients who are not participating in other clinical trials;
7. after completion of the repair, compliance with the USPHS evaluation criteria of marginal density class A cases

Exclusion Criteria:

1. obvious destruction of the apical tissue and large cysts;
2. severe periodontitis patients;
3. oral malignant tumor patients;
4. radiotherapy patients;
5. pregnant women;
6. patients with mental illness or systemic diseases;
7. people who can not take care of themselves;
8. the researchers believe that is not suitable for the test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
USPHS criteria for dental restorations assessment | 2 Years
  This criteria is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination. Some items are evaluated quantitatively, others visually.The score of all items is retained as the overall score of the restoration.

SECONDARY OUTCOMES:
Marginal Adaptation | 2 Years
  Clinical reevaluations were so far performed at baseline and 24 months after insertion according to modified United States Public Health Service (USPHS) criteria by 2 independent evaluators. A: Crown margin not discernible; probe does not catch; B: Probe catches on crown margin but no gap; gap or chipping on probing, with enamel exposed but polishable; C: Gap or chipping, with dentin or liner exposed ; D: Partial fracture, fracture, luxation.
Marginal discoloration | 2 Years
  Clinical reevaluations were so far performed at baseline and 24 months after insertion according to modified United States Public Health Service (USPHS) criteria by 2 independent evaluators. A: No discoloration on the margin between the restoration and the tooth structure; B: Superficial discoloration on the margin between the restoration and the tooth structure; does not penetrate in pulpal direction; C: Discoloration has penetrated along the margin of the restorative material in pulpal direction.
Integrity of restoration | 2 Years
  Clinical reevaluations were so far performed at baseline and 24 months after insertion according to modified United States Public Health Service (USPHS) criteria by 2 independent evaluators. A: Intact; B: Crack apparent on transillumination; C: Fracture observable; D: Crown lost(state at which interface debond occurred).

CONTACTS AND LOCATIONS:
Overall Officials: BuLing Wu, PHD, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- NanFang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun J, Ruan W, He J, Lin X, Ci B, Yin S, Yan W. Clinical efficacy of different marginal forms of endocrowns: study protocol for a randomized controlled trial. Trials. 2019 Jul 24;20(1):454. doi: 10.1186/s13063-019-3530-1. PMID 31340845